CLINICAL TRIAL: NCT01791413
Title: Effect of Pre-operative Depo Medroxyprogesterone Acetate on Serum Anti-mullerian Hormone Level After Laparoscopic Ovarian Cystectomy of Endometriomas
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Weena Krutsawad, Department of Obstetrics and Gynecology, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 02-55-13
Record Dates: First submitted 2013-02-10; First posted 2013-02-15 (Estimated); Results first posted 2013-08-23 (Estimated); Last update posted 2013-09-09 (Estimated); Status verified 2013-08

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- depot medroxyprogesterone acetate (Active Comparator)
  Interventions: Drug: depot medroxyprogesterone acetate
- No depot medroxyprogesterone acetate (No Intervention)

INTERVENTIONS:
Drug: depot medroxyprogesterone acetate — DMPA 150 mg intramuscular Before surgery 3 months (plus or minus 2 weeks)
  Arms: depot medroxyprogesterone acetate

SUMMARY:
The purpose of this study is to evaluate the ovarian reserve changes after preoperative depot medroxyprogesterone acetate (DMPA) in women with ovarian endometrioma undergoing laparoscopic cystectomy.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women 18-40 years old
* A diagnosis of endometrioma with diameter of at least 3 cm.
* Candidates for laparoscopic cystectomy

Exclusion Criteria:

* Patients' refusal to participate
* Not candidate for depot medroxyprogesterone acetate such as: cirrhosis, chronic kidney disease, venous thrombosis
* Use of estrogen-suppressive drugs in the preceding 3 months, such as:

Oral contraceptives, GnRH analogues, Progestins, Danazol

* Pathology report present no endometriosis

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2012-03; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics and Gynecology, Ratchathewi, Bangkok, Thailand

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Mar.2012-Feb.2013 University Hospital
Pre-assignment Details: Assessed for eligibility n=60 Excluded n=20 (15=not compatible with inclusion criteria 5=denied to participate)
Groups:
- Depot Medroxyprogesterone Acetate: depot medroxyprogesterone acetate : DMPA 150 mg intramuscular Before surgery 3 months (plus or minus 2 weeks)
Period: Overall Study
Arm/Group | No Depot Medroxyprogesterone Acetate | Depot Medroxyprogesterone Acetate
Started | 20 | 20
Completed | 15 | 19
Not Completed | 5 | 1
Not completed — Lost to Follow-up | 5 | 1

BASELINE CHARACTERISTICS:
Population: Lost follow up total 6 patients
Groups:
- Total: Total of all reporting groups
Arm/Group | No Depot Medroxyprogesterone Acetate | Depot Medroxyprogesterone Acetate | Total
Number analyzed (Participants) | 19 | 15 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 15 | 34
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 32.57 (5.67) | 32.46 (6.46) | 32.53 (6.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 15 | 34
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Thailand | 19 | 15 | 34

OUTCOME MEASURES:

1. Primary Outcome: Percentage Changes of Serum Anti-Mullerian Hormone (AMH) at 2-week and 3-month Post Operation
Time Frame: Within the first 2 weeks and 3 months after surgery
Measure: Median (Inter-Quartile Range); unit: percentage of serum AMH change
Groups:
- 2 wk Post op : No Depot Medroxyprogesterone Acetate: Percentage changes of serum Anti-Mullerian hormone (AMH) at 2-week post operation
- 2 wk Post op:Depot Medroxyprogesterone Acetate: depot medroxyprogesterone acetate : DMPA 150 mg intramuscular Before surgery 3 months (plus or minus 2 weeks)Percentage changes of serum Anti-Mullerian hormone (AMH) at 2-week post operation
- 3 mo. Post op: No Depot Medroxyprogesterone Acetate; 3 mo. Post op: Depot Medroxyprogesterone Acetate: Percentage changes of serum Anti-Mullerian hormone (AMH) at 3-month post operation
Arm/Group | 2 wk Post op : No Depot Medroxyprogesterone Acetate | 2 wk Post op:Depot Medroxyprogesterone Acetate | 3 mo. Post op: No Depot Medroxyprogesterone Acetate | 3 mo. Post op: Depot Medroxyprogesterone Acetate
Number analyzed (Participants) | 19 | 15 | 19 | 15
percentage of serum AMH change | -56.86 [-75.10 to -30.78] | -77.72 [-97.56 to -69.82] | -36.69 [-66.10 to -19.09] | -66.84 [-93.23 to -51.21]

ADVERSE EVENTS:
Description: serious and/or other [non-serious] adverse events were not collected/assessed
Arm/Group | DMPA
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Small sample size

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes